CLINICAL TRIAL: NCT02613195
Title: Hydrogen-Rich Celsior Solution Improve the Quality of Aging DBD Grafts in Liver/Kidney Transplantation: Prospective, Randomized Clinical Trial
Brief Title: Clinical Trial of Hydrogen-Rich Celsior Solution Applied in Aging DBD Liver/Kidney Transplantation
Acronym: HRCSDBD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RenJiH-20151020
Record Dates: First submitted 2015-10-24; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Evidence of Liver Transplantation
Keywords: Ischemia-Reperfusion Injury; oxidative stress; organ preservation; Hydrogen; Kidney Transplantation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrogen-rich Celsior solution (Experimental): Using aging liver grafts（≥60 years old)，lavaged and cold stored with hydrogen-rich Celsior solution for 2-4 hours.
  Interventions: Drug: Hydrogen-Rich Celsior Solution
- Celsior solution (No Intervention): Using aging liver/kidney grafts（≥60 years old）, lavaged and cold stored with common Celsior solution for 2-4 hours.

INTERVENTIONS:
Drug: Hydrogen-Rich Celsior Solution — Before the procedure, add hydrogen gas into Celsior solution. After harvesting the liver/kidney grafts, lavage and cold store the grafts with Hydrogen-Rich Celsior Solution.
  Other Names: HR solution
  Arms: Hydrogen-rich Celsior solution

SUMMARY:
The purpose of this study is to investigate whether hydrogen-rich Celsior solution improve the quality of aging grafts in liver/kidney transplantation.

DETAILED DESCRIPTION:
The organ shortage has been rising to impede the development of organ transplantation.To find a solution, transplantation center is working on the application of marginal grafted liver or renal, especially the aging grafts. The most common inducement of organ dysfunction during the perioperation is liver/renal ischemia-reperfusion (I/R) injury, caused by the generation of cytotoxic oxygen radicals. Hydrogen gas is a kind of reducing gas, which has been reported to display antioxidant properties and protective effects against organ dysfunction induced by various I/R injuries. Investigators will investigate whether hydrogen-rich Celsior solution improve the quality of aging grafts in liver/ kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

Donors:

1. Age of the donor ≥60 yrs.
2. The donor has no historical records of drug abuse, alcoholic abuse, homosexual,or drug addiction, etc.
3. Evaluate infections and infectious disease of the donor.
4. History of malignant tumor;
5. History of hypertension, diabetes, hemophilia, or other anticoagulant disease,kidney donor should not have a history of kidney disease.
6. Daily urine volume is approximately normal.
7. Donor should be subjected to physical examination by medical doctor of OPO stuff before donation; the OPO stuff should realize whether the potential donor has infected lesion or not, such as abscess, ulcer, lymphadenectasis， etc., and evaluate infectious risk of recipient post-operationally.
8. OPO stuff should realize the dynamic change of body temperature, as well as various intensive care parameters of the potential donor, it shall be very important to be sure whether the potential donor has pulmonary/ systemic infections or not,especially for whom has longer ICU duration (> 7 Days).
9. The potential donor should has a systolic blood pressure ≥ 50 mm Hg (1mmHg=0.133 kPa) and arterial SaO > 80%.
10. Liver Biochemistry: alanine aminotransferase (ALT) ≤ 6ULN, total bilirubin (TBil) ≤ 50umol/L;Kidney Biochemistry: serum creatinine (sCre) ≤ 2ULN;
11. Negative anti-HIV antibody;
12. Negative bacterial and fungal culture in blood;
13. Ultrasonic diagnosis of fatty liver, trauma, hematoma, lithiasis, etc., as well as size of both kidney, hydronephrosis, nephrolithiasis, etc. if possible.
14. Graft liver should be soft, normal color and even, no tumor or other abnormity;steatosis ≤ 30% by liver biopsy.Graft kidneys should have complete renal capsule with no congestion or bleeding;proximal tubular necrosis ≤ 50%, without obvious structural damage.Organ (liver and kidney) cold ischemia time (CIT) is determined as the time duration from cold preservation of organs to transplant re-perfusion. CIT of aging DBD liver and kidney graft should be ≤ 10 and16 hours, respectively.

Recipients：

1. Aged between 18-65 years old
2. MELD score ≤25,BMI≤25
3. Patients with tumor,the expected lifetime≥6 months
4. Agree to anticipate the trial and sign the informed consent

Exclusion Criteria:

* Donor's age < 60 yrs;
* The donor has historical records of drug abuse, alcoholic abuse, homosexual, or drug addiction, etc.
* The donor is HIV infected, or has severe infection, or positive bacterial and/ or fungal culture results;
* Uncontrollable hypertension, diabetics;
* Malignant tumor;
* Unstable hemodynamic response or SaO status, such as systolic pressure <50 mm Hg (1mmHg=0.133 kPa) , or arterial SaO<80%.
* Liver Biochemistry: alanine aminotransferase (ALT)>6ULN, total bilirubin (TBil)>50umol/L;
* Graft liver has a steatosis >30%, or graft kidney has a proximal tubular necrosis>50% or obvious glomerular sclerosis.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Aspartate Aminotransferase(AST)/Alanine Aminotransferase(ALT) | up to 6 months
Change From Baseline in direct bilirubin(DBil)/total bilirubin(TBil) | up to 6 months
Change From Baseline in creatinine | up to 6 months
Change From Baseline in glomerular filtration rate（GFR） | up to 6 months

SECONDARY OUTCOMES:
Pathological score of liver/kidney preservation injury during surgery | during surgery
Mitochondrial function index of hepatocyte/nephrocyte during surgery | during surgery
The total incidence of adverse events/incidence of severe adverse events | up to 6 months
postoperative complications | up to 6 months
Early graft function incidence | baseline and 6 months
Graft dysfunction incidence | baseline and 6 months
Recipient survival | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xia Qiang, investigator, Study Director — Deparment of Liver Surgery
Locations (2):
- China (2):
  - Ren Ji Hospital, Shanghai, Shanghai Municipality
  - Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai

REFERENCES:
- [Result] Abe T, Li XK, Yazawa K, Hatayama N, Xie L, Sato B, Kakuta Y, Tsutahara K, Okumi M, Tsuda H, Kaimori JY, Isaka Y, Natori M, Takahara S, Nonomura N. Hydrogen-rich University of Wisconsin solution attenuates renal cold ischemia-reperfusion injury. Transplantation. 2012 Jul 15;94(1):14-21. doi: 10.1097/TP.0b013e318255f8be. PMID 22683850
- [Result] Qian L, Shen J. Hydrogen therapy may be an effective and specific novel treatment for acute graft-versus-host disease (GVHD). J Cell Mol Med. 2013 Aug;17(8):1059-63. doi: 10.1111/jcmm.12081. Epub 2013 Jun 7. PMID 23742028
- [Result] Buchholz BM, Masutani K, Kawamura T, Peng X, Toyoda Y, Billiar TR, Bauer AJ, Nakao A. Hydrogen-enriched preservation protects the isogeneic intestinal graft and amends recipient gastric function during transplantation. Transplantation. 2011 Nov 15;92(9):985-92. doi: 10.1097/TP.0b013e318230159d. PMID 21956195
- [Result] Liu Y, Yang L, Tao K, Vizcaychipi MP, Lloyd DM, Sun X, Irwin MG, Ma D, Yu W. Protective effects of hydrogen enriched saline on liver ischemia reperfusion injury by reducing oxidative stress and HMGB1 release. BMC Gastroenterol. 2014 Jan 12;14:12. doi: 10.1186/1471-230X-14-12. PMID 24410860
- [Result] Noda K, Shigemura N, Tanaka Y, Bhama J, D'Cunha J, Kobayashi H, Luketich JD, Bermudez CA. Hydrogen preconditioning during ex vivo lung perfusion improves the quality of lung grafts in rats. Transplantation. 2014 Sep 15;98(5):499-506. doi: 10.1097/TP.0000000000000254. PMID 25121557